CLINICAL TRIAL: NCT00113880
Title: Post-Marketing Evaluation of the Safety of Influenza Virus Vaccine Live, Intranasal (FluMist) in Healthy Children and Healthy Adults 5-49 Years of Age
Brief Title: A Study to Evaluate the Safety of FluMist in Healthy Children and Healthy Adults
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: FM025
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
MeSH Terms: interventions — FluMist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 5-8 years of age, estimated to be approximately 4,000 new FluMist vaccinees per season
  Interventions: Biological: FluMist
- 2: 9-17 years of age, estimated to be approximately 5,000 new FluMist vaccinees per season
  Interventions: Biological: FluMist
- 3: 18-49 years of age, estimated to be approximately 6,000 new FluMist vaccinees per season.
  Interventions: Biological: FluMist

INTERVENTIONS:
Biological: FluMist — Nasal Sprayer dose of FluMist with annual follow up
  Groups: 1
Biological: FluMist — Nasal Sprayer dose of FluMist with annual follow up
  Groups: 2
Biological: FluMist — Nasal Sprayer dose of FluMist with annual follow up
  Groups: 3

SUMMARY:
The purpose of this study was to expand the data describing the safety profile of FluMist in the indicated populations (5-8, 9-17, and 18-49 years of age) and to assess the safety of annual revaccination in those who received FluMist in 2 or more consecutive years.

DETAILED DESCRIPTION:
The primary objective of this study was to assess the safety of FluMist vaccination by comparing the rates of medically attended events (MAEs) (including serious adverse events [SAEs], anaphylaxis, urticaria, asthma, wheezing, pre-specified grouped diagnoses, and rare events potentially related to wild-type influenza) in FluMist recipients to rates in multiple non-randomized control groups.

ELIGIBILITY:
Inclusion Criteria:

* 5-49 years of age
* Members of the Kaiser Permanente (KP) Health Care Plan within KP of Northern California, KP of Colorado, and KP of Hawaii

Exclusion Criteria:

* Must not have had any high risk underlying medical conditions, includig asthma

Ages: 5 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This is an observational study conducted over multiple years with multiple non-randomized control groups.
Sampling Method: Probability Sample
Enrollment: 63061 (Actual)
Dates: Start 2003-10; Primary Completion 2008-09 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ambrose, M.D., Study Director — MedImmune LLC
Locations (76):
- United States (76):
  - Kaiser Permanente Pediatrics, Alameda, California
  - Kaiser Permanente Pediatrics, Antioch, California
  - Kaiser Permanente Pediatrics, Clovis, California
  - Kaiser Permanente Pediatrics, Daly City, California
  - Kaiser Permanente, Davis, California
  - Kaiser Pediatric Injections, Fairfield, California
  - Kaiser Permanente-Pediatrics, Folsom, California
  - Kaiser Permanente Adult Injection, Fremont, California
  - Kaiser Permanente Pediatrics, Fremont, California
  - Kaiser Permanente Pediactrics, Fresno, California
  - Kaiser Permanente Pediatrics, Gilroy, California
  - Kaiser Pediatric Injection Station, Hayward, California
  - Kaiser Permanente, Lincoln, California
  - Kaiser Pediatric Injection Station, Livermore, California
  - Kaiser Permanente Injection Clinic, Manteca, California
  - Kaiser Permanente Pediatrics, Martinez, California
  - Kaiser Permanente Adult Medicine, Milpitas, California
  - Kaiser Permanente Employee Health, Milpitas, California
  - Kaiser Permanente Pediatrics, Milpitas, California
  - Kaiser Permanente Injection Clinic, Modesto, California
  - Kaiser Permanente Medicine Dept., Modesto, California
  - Kaiser Permanente Pediatrics, Mountain View, California
  - Kaiser Permanente Pediatrics, Napa, California
  - Kaiser Permanente Pediatrics, Novato, California
  - Kaiser Permanente Employee Health, Oakland, California
  - Kaiser Permanente Injection Clinic, Oakland, California
  - Kaiser Permanente Pediatrics, Oakland, California
  - Kaiser Permanente Regional Employee Health, Oakland, California
  - Kaiser Permanente Pediatrics, Petaluma, California
  - Kaiser Permanente Pediatrics, Pleasanton, California
  - Kaiser Permanente Pediatrics, Rancho Cordova, California
  - Kaiser Permanente, Redwood City, California
  - Kaiser Permanente Adult Injection Clinic, Richmond, California
  - Kaiser Permanente Pediatrics, Richmond, California
  - Kaiser Permanente Pediatrics, Roseville, California
  - Kaiser Permanente, Roseville, California
  - Kaiser Permanente, Point West Clinic Pediatric Injection, Sacramento, California
  - Kaiser Permanente, Sacramento, California
  - Kaiser Pediatric Injection Station, Sacramento, California
  - Kaiser Permanente Medicine Dept., Sacramento, California
  - Kaiser Permanente Medicine Dept., San Francisco, California
  - Kaiser Permanente Pediatrics, San Francisco, California
  - Kaiser Permanente Pharmacy, San Francisco, California
  - Kaiser Pediatric Adult Medicine, San Jose, California
  - Kaiser Pediatric Injection Clinic, San Jose, California
  - Kaiser Permanente Employee Health, San Rafael, California
  - Kaiser Permanente Pediatrics, San Rafael, California
  - Kaiser Permanente Adult Medicine, Santa Clara, California
  - Kaiser Permanente Employee Health, Santa Rosa, California
  - Kaiser Permanente Pediatrics, Santa Rosa, California
  - Kaiser Permanente Pediatrics, Selma, California
  - Kaiser Permanente Injection/Allergy, Stockton, California
  - Kaiser Permanente Pediatrics, Tracy, California
  - Kaiser Pediatric Injection Room, Vacaville, California
  - Kaiser Permanente Adult Medicine, Vacaville, California
  - Kaiser Permanente Injection Clinic, Vallejo, California
  - Kaiser Permanente Pediatric Injections, Vallejo, California
  - Kaiser Permanente Pediatrics, Walnut Creek, California
  - Kaiser Permanente, Hidden Lake, Arvada, Colorado
  - Kaiser Permanente, Aurora Centrepoint, Aurora, Colorado
  - Kaiser Permanente, Smoky Hill, Aurora, Colorado
  - Kaiser Permanente, Baseline, Boulder, Colorado
  - Kaiser Permanente, Boulder, Boulder, Colorado
  - Kaiser Permanente, Broomfield, Broomfield, Colorado
  - Kaiser Permanente, Skyline, Denver, Colorado
  - Kaiser Permanente, East, Denver, Colorado
  - Kaiser Permanente, Englewood, Englewood, Colorado
  - Kaiser Permanente, Highlands Ranch, Colorado
  - Kaiser Permanente, Lafayette, Colorado
  - Kaiser Permanente, Lakewood, Lakewood, Colorado
  - Kaiser Permanente Arapahoe, Littleton, Colorado
  - Kaiser Permanente, Southwest, Littleton, Colorado
  - Kaiser Permanente, Ken Caryl, Littleton, Colorado
  - Kaiser Permanente, Longmont Primary Care, Longmont, Colorado
  - Kaiser Permanente, Westminster, Westminster, Colorado
  - Kaiser Permanente, Wheatridge, Wheat Ridge, Colorado

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 5 to 49 years of age who were members of the Kaiser Permanente (KP) Health Care Plan at health care centers in Northern California, Colorado, and Hawaii. The first subject vaccinated with FluMist was on 15Oct2003 and the date of the last subject/last assessment was 30Sep2008.
Pre-assignment Details: Of 197,502 subjects, 189,174 unique subjects were included in this study, representing the total number of subjects who were defined exclusively within each season. FluMist recipients who received an additional 7,570 FluMist doses were excluded from the analysis based on the presence of high risk underlying medical conditions and other factors.
Groups:
- FluMist Recipients: Subjects who had been immunized with FluMist as part of routine clinical practice at health care centers within the KP Health Care Plan. Subjects from 5-8 years of age may have received 1 or 2 doses of FluMist, while subjects ≥ 9 years of age were expected to receive only 1 dose. FluMist recipients served as their own controls based on the observation time after vaccination. In the primary analyses using within-cohort controls, "risk" periods of Days 0 to 3 and Days 0 to 21 post vaccination were compared to "reference" observation time occurring after the respective risk periods, ie, Days 4 to 42 for the risk period of Days 0 to 3 and Days 22 to 42 for the risk period of Days 0 to 21.
- Unvaccinated Control: Non-randomized unvaccinated subjects were matched 1:1 with FluMist recipients and were selected from the pool of individuals who were members of the Kaiser Health Maintenance Organization (HMO) during the same month that the reference FluMist recipient was vaccinated, and included only those who did not receive the trivalent inactivated influenza vaccine (TIV) formulation at the Kaiser HMO. Other matching factors included age (within 1 year), gender, prior year health care utilization level (ie, similar number of hospital, emergency department (ED), and clinic visits), and medical center (only for subjects from Northern California).
- TIV-Vaccinated Control: Non-randomized TIV-vaccinated subjects matched 1:1 with FluMist recipients and were selected from the pool of individuals who received TIV but not FluMist at the Kaiser HMO during the same month that the reference FluMist recipient was vaccinated. Other matching factors included age (within 1 year), gender, prior year health care utilization level (ie, similar number of hospital, ED, and clinic visits), and medical center (only for subjects from Northern California).
Period: Overall Study
Arm/Group | FluMist Recipients | Unvaccinated Control | TIV-Vaccinated Control
Started | 63061 | 71949 | 62492
Completed | 63061 | 71949 | 62492
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluMist Recipients | Unvaccinated Control | TIV-Vaccinated Control | Total
Number analyzed (Participants) | 63061 | 71949 | 62492 | 197502
Age Continuous [Mean (Standard Deviation); unit: Years] | 17.1 (12.8) | 17.1 (12.8) | 16.8 (12.7) | 17.1 (12.8)
Gender [Number; unit: dose] — Gender data was collected per dose of intervention and not per participant and that each participant could have received more than one dose.
  dose
    Female | 41593 | 41591 | 37373 | 120557
    Male | 33116 | 33115 | 29626 | 95857

OUTCOME MEASURES:

1. Primary Outcome: Rates of Medically Attended Events (MAEs) Associated With a Significant Increased Risk in FluMist Recipients Compared to Rates in Within Cohort, Unvaccinated, and TIV Control Groups
Description: An MAE was defined as a coded medical diagnosis made by a health care provider and associated with a medical encounter (ie, a visit by a health plan member to a medical clinic or ED, or a hospital admission). Incident rate comparisons of MAEs with an identified increased risk associated with FluMist occurring in the same age group and setting across all three comparison groups, as these events are less likely to be due to chance alone.
Time Frame: 21 and 42 days
Population: Analyses were performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years). Significance was observed in the clinic setting, 21 days post Dose 1 in 7 subjects (breast lump/cyst, 9-17 yrs) and in 22 subjects (mastitis, 18-49 yrs).
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Groups:
- FluMist Recipients: Subjects who had been immunized with FluMist as part of routine clinical practice at health care centers within the Kaiser Permanente Health Care Plan. Subjects from 5-8 years of age may have received 1 or 2 doses of FluMist, while subjects ≥ 9 years of age were expected to receive only 1 dose.
- Within Cohort Control: FluMist recipients served as their own controls based on the observation time after vaccination. FluMist vaccinated cohort served as its own control. In the primary analyses using within-cohort controls, "risk" periods of Days 0 to 3 and Days 0 to 21 post vaccination were compared to "reference" observation time occurring after the respective risk periods, ie, Days 4 to 42 for the risk period of Days 0 to 3 and Days 22 to 42 for the risk period of Days 0 to 21.
- TIV-Vaccinated Control: TIV-Vaccinated Control Non-randomized TIV-vaccinated subjects matched 1:1 with FluMist recipients and were selected from the pool of individuals who received TIV but not FluMist at the Kaiser HMO during the same month that the reference FluMist recipient was vaccinated. Other matching factors included age (within 1 year), gender, prior year health care utilization level (ie, similar number of hospital, ED, and clinic visits), and medical center (only for subjects from Northern California).
Arm/Group | FluMist Recipients | Within Cohort Control | Unvaccinated Control | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 63061 | 71949 | 62492
Number analyzed (Doses) | 74709 | 74709 | 74706 | 66999
Cases per 1,000 person-months
  Breast lump/cyst | 0.33 | 0.00 | 0.00 | 0.00
  Mastitis | 1.46 | 0.61 | 0.20 | 0.23
Statistical Analysis 1: Comparison: FluMist Recipients vs Within Cohort Control; Breast lump/cyst event rates were presented per 1,000 person-months. If the control group has no event, the relative risk (RR) or hazard ratio (HR) is not estimable; Test type: Superiority or Other; p = 0.01, Exact method or Cox model — Due to the exploratory nature of the study and the lack of formal hypothesis testing, multiple confidence intervals (CIs) were constructed without multiplicity adjustment
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; Breast lump/cyst event rates were presented per 1,000 person-months. If the control group has no event, the RR or HR is not estimable; Test type: Superiority or Other; p = 0.01, Exact method or Cox model — Due to the exploratory nature of the study and the lack of formal hypothesis testing, multiple CIs were constructed without multiplicity adjustment
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.02, Exact method or Cox model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: FluMist Recipients vs Within Cohort Control; Mastitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.64 to 3.92]
Statistical Analysis 5: Comparison: FluMist Recipients vs Unvaccinated Control; Mastitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 7.35, 95% CI 2-sided [2.20 to 24.54]
Statistical Analysis 6: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Mastitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 7.17, 95% CI 2-sided [2.13 to 24.13]

2. Primary Outcome: Rates of MAEs Associated With a Significant Decreased Risk in FluMist Group Compared to Rates in Within Cohort, Unvaccinated, and TIV Control Groups
Description: Incident rate comparisons of MAEs with an identified decreased risk associated with FluMist occuring in the same age group and setting across all three comparison groups, as these events are less likely to be due to chance alone. All terms were analyzed for the entire population regardless of gender.
Time Frame: 21 and 42 days
Population: Analyses performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (1 or 2 for ages 5-8 years). Significance observed in the clinic, 21 days post Dose 1 in 1 subj. (heart murmur, all ages combined); 18 and 19 subj.(pregnancy exam, 18-49 and all ages combined).
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Within Cohort Control | Unvaccinated Control | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 63061 | 71949 | 62492
Number analyzed (Doses) | 74709 | 74709 | 74706 | 66999
Cases per 1,000 person-months
  Heart murmur | 0.02 | 0.16 | 0.15 | 0.21
  Pregnancy exam, 18-49 yrs | 1.19 | 3.06 | 23.48 | 70.41
  Pregnancy exam, all ages combined | 0.37 | 0.89 | 7.18 | 20.09
Statistical Analysis 1: Comparison: FluMist Recipients vs Within Cohort Control; Heart murmur event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.03, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.05, 95% CI 2-sided [0.00 to 0.79]
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; Heart murmur event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.05, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.02 to 1.00]
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Heart murmur event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.11, 95% CI 2-sided [0.01 to 0.86]
Statistical Analysis 4: Comparison: FluMist Recipients vs Within Cohort Control; Pregnancy exam/supervision event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.20 to 0.70] — Population was the 18-49 year age group
Statistical Analysis 5: Comparison: FluMist Recipients vs Within Cohort Control; Pregnancy exam/supervision event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.22 to 0.74] — Population was the all ages combined group
Statistical Analysis 6: Comparison: FluMist Recipients vs Unvaccinated Control; Pregnancy exam/supervision event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.05, 95% CI 2-sided [0.03 to 0.08] — Population was the 18-49 year age and the all ages combined groups
Statistical Analysis 7: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Pregnancy exam/supervision event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox; Hazard Ratio (HR) = 0.02, 95% CI 2-sided [0.01 to 0.03] — Population was the 18-49 year age and all ages combined groups

3. Primary Outcome: Rates of Anaphylaxis and Urticaria in FluMist Recipients Compared to Rates in Within Cohort, Unvaccinated, and TIV Control Groups
Description: Incident rate comparisons associated with a significantly increased risk in FluMist recipients compared to the within cohort control group for urticaria; there was no increased risk compared to the unvaccinated and TIV control groups and there were no anaphylaxis events that occurred within the 3-day risk period post vaccination.
Time Frame: 3 days
Population: Analyses were performed by period (3 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years).
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Within Cohort Control | Unvaccinated Control | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 63061 | 71949 | 62492
Number analyzed (Doses) | 74709 | 74709 | 74706 | 66999
Cases per 1,000 person-months | 1.19 | 0.89 | 0.83 | 1.58
Statistical Analysis 1: Comparison: FluMist Recipients vs Within Cohort Control; Urticaria event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 2.06, 95% CI 2-sided [1.02 to 4.13]

4. Primary Outcome: Rates of MAEs Within the Pre-specified Grouped Diagnoses In The FluMist Group Compared to Rates in Within Cohort, Unvaccinated, and TIV Control Groups.
Description: There were no acute respiratory tract events, acute gastrointestinal tract events, or systemic bacterial infections with an identified increased or decreased risk associated with FluMist occuring in the same age group and setting across all three comparison groups.
Time Frame: 21 and 42 days
Population: Analyses were performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years).
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Within Cohort Control | Unvaccinated Control | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 63061 | 71949 | 62492
Number analyzed (Doses) | 74709 | 74709 | 74706 | 66999
Cases per 1,000 person-months | 0 | 0 | 0 | 0

5. Primary Outcome: Rates of Asthma and Wheezing Within 21 and 42 Days in FluMist Recipients Compared to Rates in the Within Cohort and Unvaccinated Control Groups
Description: Incident rate comparisons associated with a significantly decreased risk in FluMist recipients compared to the within cohort control observed for all ages and 5-8 years of age within 21 days and compared to the unvaccinated control obseved for 18-49 years of age within 42 days. No asthma and wheezing incidence rate comparisons were significantly increased in FluMist recipients compared to the within cohort or unvaccinated control groups.
Time Frame: 21 and 42 days
Population: Analyses were performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years). Significance was observed across all settings, post Dose 1 within 21 days for within cohort and within 42 days for unvaccinated.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Within Cohort Control | Unvaccinated Control
Number analyzed (Participants) | 63061 | 63061 | 71949
Number analyzed (Doses) | 74709 | 74709 | 74706
Cases per 1,000 person-months
  Any asthma or wheezing event, all ages, 21 d | 2.42 | 3.42 | 2.52
  Any asthma or wheezing event, 21 d, 5-8 | 3.28 | 5.59 | 3.03
  Any asthma or wheezing event, 42 d, 18-49 | 1.48 | NA — No data for this timepoint | 2.18
Statistical Analysis 1: Comparison: FluMist Recipients vs Within Cohort Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.56 to 0.89] — Population: all ages combined within 21 days. The rate of events during the risk period represents the numerator; the rate of events during the control period represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs Within Cohort Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.59, 95% CI 2-sided [0.41 to 0.83] — Population: 5-8 years within 21 days. The rate of events during the risk period represents the numerator; the rate of events during the control period represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs Unvaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.68, 95% CI 2-sided [0.46 to 0.99] — Population: 18-49 years within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in unvaccinated controls represents the denominator

6. Primary Outcome: Rates of Asthma and Wheezing Within 21 and 42 Days in FluMist Recipients Compared to Rates in the TIV Control Group
Description: Incident rate comparisons associated with a significantly decreased risk in FluMist recipients compared to the TIV control group for all ages, 5-8, 9-17, and 18-49 years of age. No asthma and wheezing incidence rate comparisons were significantly increased in FluMist recipients compared to the TIV control group.
Time Frame: 21 and 42 days
Population: Analyses were performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years). Significance was observed across all settings, post Dose 1 within 21 days and 42 days (all age groups) and post Dose 2 (PD2) within 42 days (5-8 yrs).
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Any asthma or wheezing event, 21 d, all ages | 2.30 | 3.20
  Any asthma or wheezing event, 21 d, 5-8 | 3.07 | 10.07
  Any asthma or wheezing event, 21 d, 9-17 | 2.43 | 7.15
  Any asthma or wheezing event, 21 d, 18-49 | 1.24 | 2.94
  Any asthma or wheezing event, 42 d, all ages | 2.76 | 7.23
  Any asthma or wheezing event, 42 d, 5-8 | 4.11 | 10.28
  Any asthma or wheezing event, 42 d, 9-17 | 2.70 | 7.57
  Any asthma or wheezing event, 42 d, 18-49 | 1.37 | 3.37
  Any asthma or wheezing event, 42 d, PD2, 5-8 | 7.10 | 14.99
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.33, 95% CI 2-sided [0.27 to 0.41] — Population: all ages combined within 21 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.30, 95% CI 2-sided [0.22 to 0.42] — Population: 5-8 years within 21 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.34, 95% CI 2-sided [0.24 to 0.47] — Population: 9-17 years within 21 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.42, 95% CI 2-sided [0.23 to 0.75] — Population: 18-49 years within 21 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 5: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.38, 95% CI 2-sided [0.33 to 0.44] — Population: all ages combined within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 6: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.40, 95% CI 2-sided [0.32 to 0.50] — Population: 5-8 years within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 7: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.36, 95% CI 2-sided [0.28 to 0.45] — Population: 9-17 years within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 8: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.41, 95% CI 2-sided [0.27 to 0.60] — Population: 18-49 years within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 9: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.05, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.21 to 0.99] — Population: 5-8 years, PD2 within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator

7. Primary Outcome: Rates of Asthma and Wheezing Within 180 Days in FluMist Recipients Compared to Rates in the Unvaccinated Control Group
Description: Incident rate comparisons associated with a significantly decreased risk in FluMist recipients compared to the unvaccinated control group for all ages, 5-8, and 9-17 years of age. No asthma and wheezing incidence rate comparisons were significantly increased in FluMist recipients compared to the unvaccinated control group.
Time Frame: 180 days
Population: Analyses performed by period (180 days), age group (5-8, 9-17, 18-49 yrs), setting (clinic, hospital, or ED), and number of doses (1 or 2 for 5-8 yrs). Significance was observed for asthma/reactive airway disease (RAD) and any ashtma or wheezing event across all settings, PD1 (all ages and 9-17 yrs) and PD2 (5-8 yrs).
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Unvaccinated Control
Number analyzed (Participants) | 63061 | 71949
Number analyzed (Doses) | 74709 | 74706
Cases per 1,000 person-months
  Any asthma or wheezing event, PD1, all ages | 4.07 | 4.45
  Any asthma or wheezing event, PD1, 9-17 | 4.00 | 4.81
  Asthma/RAD, PD1, all ages | 3.04 | 3.48
  Asthma/RAD, PD1, 9-17 | 3.10 | 3.94
  Asthma/RAD, PD2, 5-8 | 2.69 | 5.54
Statistical Analysis 1: Comparison: FluMist Recipients vs Unvaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.86 to 0.98] — Population: all ages combined, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.75 to 0.92] — Population: 9-17 yrs., within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs Unvaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.81 to 0.94] — Population: All ages, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs Unvaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.70 to 0.88] — Population: 9-17 yrs, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 5: Comparison: FluMist Recipients vs Unvaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.29 to 0.79] — Population: 5-8yrs, within 180 days, PD2. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator

8. Primary Outcome: Rates of Asthma and Wheezing Within 180 Days in FluMist Recipients Compared to Rates in the TIV Control Group
Description: as for outcome 6
Time Frame: 180 days
Population: Analyses performed by period (180 days), age group (5-8, 9-17, 18-49 yrs), setting (clinic, hospital, or ED), and number of doses (1 or 2 for 5-8 yrs). Significance was observed for asthma/RAD, wheezing/shortness of breath (SOB), and any ashtma or wheezing event across all settings, PD1 (all age groups) and PD2.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Any asthma or wheezing event, PD1, all ages | 4.06 | 8.50
  Any asthma or wheezing event, PD1, 5-8 | 5.88 | 11.45
  Any asthma or wheezing event, PD1, 9-17 | 3.96 | 9.41
  Any asthma or wheezing event, PD1, 18-49 | 2.27 | 3.98
  Any asthma or wheezing event, PD2, 5-8 | 5.76 | 11.40
  Asthma/RAD, PD1, all ages | 3.04 | 7.23
  Asthma/RAD, PD1, 5-8 | 3.87 | 9.14
  Asthma/RAD, PD1, 9-17 | 3.08 | 8.25
  Asthma/RAD, PD1, 18-49 | 2.10 | 3.65
  Asthma/RAD, PD2, 5-8 | 2.18 | 7.67
  Wheezing/SOB, PD1, all ages | 1.15 | 1.53
  Wheezing/SOB, PD1, 5-8 | 2.29 | 2.77
  Wheezing/SOB, PD1, 9-17 | 0.98 | 1.37
  Wheezing/SOB, PD1, 18-49 | 0.19 | 0.41
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.48, 95% CI 2-sided [0.45 to 0.51] — Population: all ages combined, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.51, 95% CI 2-sided [0.47 to 0.56] — Population: 5-8 yrs, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.42, 95% CI 2-sided [0.38 to 0.46] — Population: 9-17 yrs, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.57, 95% CI 2-sided [0.49 to 0.67] — Population: 18-49yrs, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 5: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.51, 95% CI 2-sided [0.33 to 0.76] — Population: 5-8 yrs, within 180 days, PD2. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 6: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.42, 95% CI 2-sided [0.39 to 0.45] — Population: all ages, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 7: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.42, 95% CI 2-sided [0.38 to 0.47] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 8: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.37, 95% CI 2-sided [0.34 to 0.41] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 9: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.05, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.49 to 0.68] — Population: 18-49 yrs, within 180 days, PD1. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 10: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/Rad event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Difference (RD) = 0.28, 95% CI 2-sided [0.15 to 0.52] — [estimate comment as in outcome 8, analysis 5]
Statistical Analysis 11: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Wheezing/SOB event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.66 to 0.85] — [estimate comment as in outcome 8, analysis 6]
Statistical Analysis 12: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Wheezing/SOB event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.83, 95% CI 2-sided [0.70 to 0.97] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 13: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Wheezing/SOB event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.72, 95% CI 2-sided [0.58 to 0.88] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 14: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Wheezing/SOB event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.27 to 0.78] — [estimate comment as in outcome 8, analysis 9]

9. Primary Outcome: Rare Events Potentially Related to Wild-type Influenza in FluMist Recipients Compared to TIV and Unvaccinated Control Groups
Description: Incident rate comparisons associated with a significantly decreased risk in FluMist recipients compared to TIV controls; there was no significantly decreased risk compared to the within cohort and unvaccinated controls. No MAEs potentially related to wild-type influenza were associated with a significantly increased risk in FluMist recipients.
Time Frame: 21 and 42 days
Population: Analyses were performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years). significance was observed for encephalitis/encephalopathy, for all age groups, across all settings within 42 days, PD1.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Groups:
- Unvaccinated Controls: Non-randomized unvaccinated subjects were matched 1:1 with FluMist recipients and were selected from the pool of individuals who were members of the Kaiser Health Maintenance Organization (HMO) during the same month that the reference FluMist recipient was vaccinated, and included only those who did not receive the trivalent inactivated influenza vaccine (TIV) formulation at the Kaiser HMO. Other matching factors included age (within 1 year), gender, prior year health care utilization level (ie, similar number of hospital, emergency department (ED), and clinic visits), and medical center (only for subjects from Northern California).
Arm/Group | FluMist Recipients | TIV-Vaccinated Control | Unvaccinated Controls
Number analyzed (Participants) | 63061 | 62492 | 71949
Number analyzed (Doses) | 74709 | 66999 | 74706
Cases per 1,000 person-months | 0.00 | 0.05 | 0.00
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Encephalitis/encephalopathy event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.00, 95% CI 2-sided [0.00 to 0.82] — The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator

10. Primary Outcome: Rates of Serious Adverse Events (SAEs) in FluMist Recipients Compared to Rates in Unvaccinated Control Group
Description: Incident rate comparisons of SAEs with an identified decreased risk associated with FluMist compared to unvaccinated controls; no decreased risk was observed in compariosn to the within cohort control. There were no SAE incidence rate comparisons that were significantly increased in FluMist recipients.
Time Frame: 21 and 42 days
Population: Analyses were performed by period (21 and 42 days), age group (5-8, 9-17, 18-49 years of age), setting (clinic, hospital, or ED), and number of doses (one or two for ages 5-8 years). Significance was observed in the any/death setting, 21 and 42 days post Dose 1, for all ages and 18-49.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Unvaccinated Control
Number analyzed (Participants) | 63061 | 71949
Number analyzed (Doses) | 74709 | 74706
Cases per 1,000 person-months
  Any SAE, all ages, 21 days | 1.12 | 1.72
  Any SAE, 18-49, 21 days | 1.33 | 3.85
  Any SAE, all ages, 42 days | 0.98 | 1.64
  Any SAE, 18-49, 42 days | 1.28 | 3.87
Statistical Analysis 1: Comparison: FluMist Recipients vs Unvaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.47 to 0.91] — Population: all ages, within 21 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.21 to 0.57] — Population: 18-49 yrs, within 21 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs Unvaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.47 to 0.77] — Population: all ages, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs Unvaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.23 to 0.48] — Population: 18-49 yrs, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator

11. Primary Outcome: Rates of SAEs in FluMist Recipients Compared to Rates in TIV Controls
Description: Incident rate comparisons of SAEs with an identified decreased risk associated with FluMist compared to TIV controls. There were no SAE incidence rate comparisons that were significantly increased in FluMist recipients.
Time Frame: 21 and 42 days
Population: as for outcome 10
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Any SAE, all ages, 21 days | 1.12 | 0.00
  Any SAE, 18-49, 21 days | 1.33 | 0.00
  Any SAE, all ages, 42 days | 0.98 | 0.23
  Any SAE, 18-49, 42 days | 1.28 | 0.23
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.47 to 0.91] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.21 to 0.57] — [estimate comment as in outcome 10, analysis 2]
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.47 to 0.77] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 4: Comparison: FluMist Recipients vs TIV-Vaccinated Control; SAE event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.23 to 0.48] — [estimate comment as in outcome 10, analysis 4]

12. Primary Outcome: Rates of Hospitalizations and Deaths Within 180 Days in FluMist Recipients Compared to Rates in Unvaccinated Controls
Description: Incident rate comparisons of hospitalizations and deaths with an identified decreased risk associated with FluMist compared to unvaccinated controls. There were no hospitalization or death incidence rate comparisons that were significantly increased in FluMist recipients.
Time Frame: 180 days
Population: Analyses were performed by period (180 days), age group (5-8, 9-17, 18-49 years of age), and number of doses (one or two for ages 5-8 years). Significance was observed in the hospitalization/death setting, 180 days post Dose 1, for all ages and 18-49.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Unvaccinated Control
Number analyzed (Participants) | 63061 | 71949
Number analyzed (Doses) | 74709 | 74706
Cases per 1,000 person-months
  Any hosp. or death, all ages | 0.97 | 1.49
  Any hosp. or death, 18-49 | 1.46 | 3.36
Statistical Analysis 1: Comparison: FluMist Recipients vs Unvaccinated Control; Hospitalization or death event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.57 to 0.73] — Population: all ages, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; Hospitalization or death event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.36 to 0.51] — Population: 18-49 yrs, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator

13. Primary Outcome: Rates of Hospitalizations and Deaths Within 180 Days in FluMist Recipients Compared to Rates in TIV Controls
Description: Incident rate comparisons of hospitalizations and deaths with an identified decreased risk associated with FluMist compared to TIV controls. There were no hospitalization or death incidence rate comparisons that were significantly increased in FluMist recipients.
Time Frame: 180 days
Population: Analyses were performed by period (180 days), age group (5-8, 9-17, 18-49 years of age), and number of doses (one or two for ages 5-8 years). Significance was observed in the hospital/death setting 180 days post Dose 1, for all ages and 18-49.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Any hosp or death, all ages | 0.95 | 3.12
  Any hosp or death, 18-49 | 1.46 | 9.10
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Hospitalization or death event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.26 to 0.33] — Population: all ages, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Hospitalization or death event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.13 to 0.18] — Population: 18-49 yrs, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator

14. Secondary Outcome: Rates of MAEs Associated With a Significant Decreased Risk in the Subset of Individuals Who Received FluMist in 2 or More Consecutive Years Compared to Rates in Within Cohort Controls
Description: Incident rate comparisons of MAEs with an identified decreased risk in FluMist recipients receiving FluMist in 2 or more consecutive seasons compared to rates in within cohort controls within 21 days. There was no significant decreased risk in comparison to unvaccinated or TIV controls within the 21-day timeframe.
Time Frame: 21 days
Population: Analyses performed by period (3, 21, and 42 days), age group (5-8, 9-17, 18-49 years of age), and setting (clinic, hospital, or ED), post Doe 1. FluMist recipients who were part of the main analysis and received FluMist in both the current and the immediate prior season(s) were included in this analysis. Significance observed across all settings.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Within Cohort Control
Number analyzed (Participants) | 63061 | 63061
Number analyzed (Doses) | 74709 | 74709
Cases per 1,000 person-months
  Sinusitis, 18-49 | 2.57 | 7.03
  URI, all ages | 10.24 | 14.79
  URI, 9-17 | 19 | 38
  URI, 9-17 | 7.26 | 14.90
  URI, 18-49 | 11.16 | 15.86
  Any acute resp. tract event, all ages | 29.20 | 37.45
  Any acute resp. tract event , 9-17 | 23.03 | 33.15
  Any acute resp. tract event ,18-49 | 21.54 | 30.09
Statistical Analysis 1: Comparison: FluMist Recipients vs Within Cohort Control; Sinusitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.16, 95% CI 2-sided [0.03 to 0.93] — Population: 18-49 within 21 days. The rate of events during the risk period represents the numerator; the rate of events during the control period represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs Within Cohort Control; URI event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.40 to 0.92] — Population: all ages, within 21 days. The rate of events during the risk period represents the numerator; the rate of events during the control period represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs Within Cohort Control; URI event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.28 to 0.84] — Population: 9-17 years, within 21 days. The rate of events during the risk period represents the numerator; the rate of events during the control period represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs Within Cohort Control; URI event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.10 to 0.78] — Population: 18-49 years, within 21 days. The rate of events during the risk period represents the numerator; the rate of events during the control period represents the denominator
Statistical Analysis 5: Comparison: FluMist Recipients vs Within Cohort Control; Any acute resp. tract event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.63 to 0.96] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 6: Comparison: FluMist Recipients vs Within Cohort Control; Any acute resp. tract event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.03, Fisher Exact — [p-value comment as in outcome 1, analysis 2]; Risk Ratio (RR) = 0.69, 95% CI 2-sided [0.50 to 0.97] — [estimate comment as in outcome 14, analysis 3]
Statistical Analysis 7: Comparison: FluMist Recipients vs Within Cohort Control; Any acute resp. tract event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.41, 95% CI [0.21 to 0.79] — [estimate comment as in outcome 14, analysis 4]

15. Secondary Outcome: Rates of MAEs Associated With a Significant Increased Risk in the Subset of Individuals Who Received FluMist in 2 or More Consecutive Years Compared to Rates in Unvaccinated Controls
Description: Incident rate comparisons of MAEs with an identified increased risk in FluMist recipients receiving FluMist in 2 or more consecutive seasons compared to rates in unvaccinated recipients. There was no increased risk at 3 or 21 days and there was no increased risk compared to the Within Cohort or TIV control groups.
Time Frame: 42 days
Population: as for outcome 14
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Unvaccinated Control
Number analyzed (Participants) | 63061 | 71949
Number analyzed (Doses) | 74709 | 74706
Cases per 1,000 person-months
  Sinusitis, all ages, 42 days | 3.74 | 1.92
  IBS, all ages, 42 days | 0.57 | 0.77
Statistical Analysis 1: Comparison: FluMist Recipients vs Unvaccinated Control; Sinusitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.95, 95% CI 2-sided [1.14 to 3.34] — [estimate comment as in outcome 10, analysis 3]
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; Irritable bowel syndrome event rates were presented per 1,000 person-months. If the control group has no event, the RR or HR is not estimable; Test type: Superiority or Other; p = 0.02, Exact method or Cox model — [p-value comment as in outcome 1, analysis 2]

16. Secondary Outcome: Rates of MAEs Associated With a Significant Decreased Risk in the Subset of Individuals Who Received FluMist in 2 or More Consecutive Years Compared to Rates in TIV Controls Within 42 Days
Description: Incident rate comparisons of MAEs with an identified decreased risk in FluMist recipients receiving FluMist in 2 or more consecutive seasons compared to rates in TIV recipients within 42 days. There was no significant decreased risk in comparison to unvaccinated controls within the 42-day timeframe.
Time Frame: 42 days
Population: as for outcome 14
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Asthma/RAD, all ages | 1.22 | 3.87
  Asthma/RAD, 5-8 | 1.82 | 5.11
  Asthma/RAD, 9-17 | 1.43 | 4.28
  Pharyngitis, all ages | 8.18 | 11.06
  Pharyngitis, 18-49 | 2.77 | 7.42
  Any acute resp. tract event, all ages | 30.72 | 36.86
  Any acute resp. tract event , 9-17 | 24.81 | 34.06
  Any asthma or wheezing event, all ages | 2.04 | 5.31
  Any asthma or wheezing event, 9-17 | 2.04 | 5.92
  Any asthma or wheezing event,18-49 | 0.00 | 2.31
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.15 to 0.57] — Population: all ages, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.03, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.12 to 0.92] — Population: 5-8, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.13 to 0.74] — Population: 9-17, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Pharyngitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.55 to 0.99] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 5: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Pharyngitis event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.04, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.14 to 0.93] — Population: 18-49 years, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 6: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any acute respiratory tract event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.71 to 0.97] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 7: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any acute respiratory tract event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.92] — [estimate comment as in outcome 16, analysis 3]
Statistical Analysis 8: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.22 to 0.61] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 9: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.16 to 0.68] — [estimate comment as in outcome 16, analysis 3]
Statistical Analysis 10: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.03, Fisher Exact; Risk Ratio (RR) = 0.00, 95% CI 2-sided [0.00 to 0.82] — Population: 18-49, within 42 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator

17. Secondary Outcome: Rates of MAEs Associated With a Significant Decreased Risk Within 180 Days in the Subset of Individuals Who Received FluMist in 2 or More Consecutive Years Compared to Rates in Unvaccinated Controls
Description: Incident rate comparisons of MAEs within 180 days with an identified decreased risk associated with FluMist recipients compared to Unvaccinated Controls. There were no MAE incidence rate comparisons that were significantly increased in FluMist recipients compared to Unvaccinated Controls.
Time Frame: 180 days
Population: Analyses performed by period (180 days), age group (5-8, 9-17, 18-49 years of age), and setting (clinic, hospital, or ED), post Doe 1. FluMist recipients who were part of the main analysis and received FluMist in both the current and the immediate prior season(s) were included in this analysis. Significance observed across all settings.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | Unvaccinated Control
Number analyzed (Participants) | 63061 | 71949
Number analyzed (Doses) | 74709 | 74706
Cases per 1,000 person-months
  Asthma/RAD, all ages | 2.88 | 3.98
  Asthma/RAD, 9-17 | 3.11 | 4.63
  Any asthma or wheezing event, all ages | 3.70 | 4.93
  Any asthma or wheezing event, 9-17 | 3.80 | 5.25
Statistical Analysis 1: Comparison: FluMist Recipients vs Unvaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.91] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: FluMist Recipients vs Unvaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.49 to 0.91] — Population: 9-17 years, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the unvaccinated controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs Unvaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.61 to 0.92] — [estimate comment as in outcome 12, analysis 1]
Statistical Analysis 4: Comparison: FluMist Recipients vs Unvaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.52 to 0.91] — [estimate comment as in outcome 17, analysis 2]

18. Secondary Outcome: Rates of MAEs Associated With a Significant Decreased Risk Within 180 Days in the Subset of Individuals Who Received FluMist in 2 or More Consecutive Years Compared to Rates in TIV Controls
Description: Incident rate comparisons of MAEs within 180 days with an identified decreased risk associated with FluMist recipients compared to TIV recipients. There were no MAE incidence rate comparisons that were significantly increased in FluMist recipients compared to TIV recipients.
Time Frame: 180 days
Population: as for outcome 17
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Asthma/RAD, all ages | 2.80 | 6.77
  Asthma/RAD, 5-8 | 3.19 | 8.49
  Asthma/RAD, 9-17 | 3.09 | 7.37
  Asthma/RAD, 18-49 | 1.64 | 3.29
  Any asthma or wheezing event, all ages | 3.62 | 7.95
  Any asthma or wheezing event, 5-8 | 4.86 | 9.94
  Any asthma or wheezing event, 9-17 | 3.82 | 8.83
  Any asthma or wheezing event,18-49 | 1.64 | 3.51
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.33 to 0.51] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.26 to 0.55] — Population: 5-8 years, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 3: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.31 to 0.56] — Population: 9-17 years, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 4: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Asthma/RAD event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.02, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.26 to 0.91] — Population: 18-49 years, within 180 days. The rate of events in FluMist recipients represents the numerator; the rate of events in the TIV controls represents the denominator
Statistical Analysis 5: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.45, 95% CI [0.37 to 0.55] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.35 to 0.67] — [estimate comment as in outcome 18, analysis 2]
Statistical Analysis 7: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.33 to 0.56] — [estimate comment as in outcome 18, analysis 3]
Statistical Analysis 8: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Any asthma or wheezing event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.25 to 0.85] — [estimate comment as in outcome 18, analysis 4]

19. Secondary Outcome: Rates of SAEs and Hospitalizations or Deaths Within 180 Days in the Subset of Individuals Who Received FluMist in 2 or More Consecutive Years Compared to Rates in Unvaccinated and TIV Controls
Description: Incident rate comparisons of SAEs and hospitalizations or deaths with an identified decreased risk associated with FluMist recipients compared to TIV recipients; there were no significant decreases compared to the unvaccinated controls. There were no SAE and hospitalization or death incidence rate comparisons that were significantly increased in FluMist recipients compared to their controls.
Time Frame: 180 days
Population: Analyses were performed by period (180 days) and age group (5-8, 9-17, 18-49 years of age), post Dose 1. recipients who were part of the main analysis and received FluMist in both the current and the immediate prior season(s) were included in this analysis. Significance was observed for any hospitalization or death, for all ages and 18-49.
Measure: Number; unit: Cases per 1,000 person-months
Units Other Than Participants: Doses
Arm/Group | FluMist Recipients | TIV-Vaccinated Control
Number analyzed (Participants) | 63061 | 62492
Number analyzed (Doses) | 74709 | 66999
Cases per 1,000 person-months
  Any hosp or death, all ages | 0.91 | 1.93
  Any hosp or death, 18-49 | 1.75 | 5.50
Statistical Analysis 1: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Hospitalization or death event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.32 to 0.69] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: FluMist Recipients vs TIV-Vaccinated Control; Hospitalization or death event rates were presented per 1,000 person-months; Test type: Superiority or Other; p = 0.01, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.17 to 0.54] — [estimate comment as in outcome 13, analysis 2]

20. Secondary Outcome: Rates of Solicited Adverse Events in Subsets of FluMist Recipients During the First Year of the Trial (2003-2004 Influenza Season)
Time Frame: Within 2-3 days of vaccination
Population: Subsets of FluMist recipients 5-8, 9-17, and 18-49 years of age
Measure: Number; unit: Percentage of FluMist recipients
Groups:
- FluMist Recipients (5-8 Years Old): Subjects who had been immunized with FluMist as part of routine clinical practice at health care centers within the Kaiser Permanente Health Care Plan. Subjects from 5-8 years of age may have received 1 or 2 doses of FluMist.
- FluMist Recipients (9-17 Years Old); FluMist Recipients (18-49 Years Old): Subjects who had been immunized with FluMist as part of routine clinical practice at health care centers within the Kaiser Permanente Health Care Plan. Subjects ≥ 9 years of age were expected to receive only 1 dose.
Arm/Group | FluMist Recipients (5-8 Years Old) | FluMist Recipients (9-17 Years Old) | FluMist Recipients (18-49 Years Old)
Number analyzed (Participants) | 749 | 683 | 643
Percentage of FluMist recipients
  Fever | 8.3 | 6.1 | 6.8
  Runny nose | 34.3 | 30.3 | 41.7
  Cough | 17.6 | 11.4 | 13.1
  Sore throat | 9.5 | 9.0 | 20.9
  Irritability | 5.9 | 4.4 | 6.8
  Headache | 9.2 | 15.2 | 21.7
  Chillls | 3.6 | 4.2 | 7.8
  Vomiting | 2.3 | 1.3 | 0.8
  Muscle aches | 4.3 | 5.2 | 12.7
  Fatigue | 10.8 | 12.9 | 18.1

21. Secondary Outcome: Rates of Solicited Adverse Events in Subsets of FluMist Recipients During the First Year of the Trial (2003-2004 Influenza Season)
Time Frame: Within 14 days of vaccination
Population: Subsets of FluMist recipients 5-8, 9-17, and 18-49 years of age
Measure: Number; unit: Percentage of FluMist recipients
Arm/Group | FluMist Recipients (5-8 Years Old) | FluMist Recipients (9-17 Years Old) | FluMist Recipients (18-49 Years Old)
Number analyzed (Participants) | 749 | 683 | 643
Percentage of FluMist recipients
  Fever | 13.4 | 11.0 | 7.7
  Runny nose | 38.2 | 33.4 | 38.6
  Cough | 25.6 | 18.8 | 17.3
  Sore throat | 15.8 | 17.4 | 20.3
  Irritability | 8.6 | 5.6 | 7.2
  Headache | 11.0 | 22.2 | 26.8
  Chillls | 5.5 | 7.2 | 10.0
  Vomiting | 5.7 | 4.1 | 1.6
  Muscle aches | 8.4 | 9.0 | 16.8
  Fatigue | 12.4 | 15.0 | 18.6

ADVERSE EVENTS:
Time Frame: 3, 21, 42 days, and 6 months post vaccination
Description: This study assessed for medically attended events (MAEs) not adverse events. An MAE was defined as a coded medical diagnosis made by a health care provider and associated with a medical encounter (ie, a visit by a health plan member to a medical clinic or ED, or a hospital admission. Results for MAEs are reported in the Outcome Measures.
Arm/Group | FluMist Recipients
Serious Adverse Events (participants affected / at risk) | 202/63061
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluMist Recipients (N=63061)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Cleft palate (Congenital, familial and genetic disorders) | 1 (1)
Congenital anomaly (Congenital, familial and genetic disorders) | 3 (3)
Eye anterior chamber congenital anomaly (Congenital, familial and genetic disorders) | 1 (1)
Factor ix deficiency (Congenital, familial and genetic disorders) | 1 (1)
Pierre robin syndrome (Congenital, familial and genetic disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2)
Goitre (Endocrine disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Colitis ulcerative (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Malocclusion (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (4)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 4 (4)
Abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 9 (9)
Arthritis bacterial (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Psoas abscess (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 15 (15)
Open wound (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Autism (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 6 (6)
Febrile convulsion (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hemicephalalgia (Nervous system disorders) | 1 (1)
Meningitis eosinophilic (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1)
Viith nerve paralysis (Nervous system disorders) | 4 (4)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 8 (8)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1)
Anorexia nervosa (Psychiatric disorders) | 1 (1)
Dependence (Psychiatric disorders) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 15 (15)
Suicide attempt (Psychiatric disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Elective procedure (Surgical and medical procedures) | 2 (2)
Female sterilisation (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Kawasaki's disease (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.